CLINICAL TRIAL: NCT03794193
Title: The Effect of Unfavorable Histological Features on the Oncological Outcomes of Colon Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Chinese Academy of Medical Sciences (Other); West China Hospital (Other); Sixth Affiliated Hospital, Sun Yat-sen University (Other); Peking University First Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: ZS-1653
Record Dates: First submitted 2018-09-09; First posted 2019-01-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Radical resection of colon cancer — The patients with colon cancer will receive radical surgery. Adjuvant chemotherapy will be given according to the results of postoperative histological results.
  Other Names: Chemotherapy

SUMMARY:
To explore the effect of unfavorable histological features on the clinical outcomes of patients receiving radical resection of colon cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-100 years old;
2. Postoperative pathology confirmed colon adenocarcinoma;
3. The tumor is located from the cecum to the sigmoid colon;
4. No distant organ metastasis;

Exclusion Criteria:

1. Simultaneous or metachronous multiple primary colorectal cancer;
2. History of previous malignant tumors (except for completely cured cervical carcinoma in situ or basal cell carcinoma or squamous epithelial skin cancer)
3. local excision procedure;
4. palliative resection (R2 resection);
5. pregnant or lactating women.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Colon cancer patients with or without unfavorable histological features
Sampling Method: Probability Sample
Enrollment: 1367 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
3-year Disease-free Survival | Within 3 years after surgery
  The time from the time of surgery to the time of recurrence or death from any cause, calculated on a monthly basis, with the most recent recurrence and metastasis.

SECONDARY OUTCOMES:
3-year Over-all Survival | Within 3 years after surgery
  The time from the time of surgery to the time of recurrence or death from any cause, calculated on a monthly basis.
Postoperative complication rate | Within 30 days after surgery
Postoperative mortality rate | Within 30 days after surgery
Local recurrence rate | Within 3 years after surgery
Distant organ metastasis rate | Within 3 years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yi Xiao, MD, Principal Investigator — Peking Union Medical College Hospital

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data can be shared with all researchers involved in the study.

REFERENCES:
- [Derived] Li K, Zhao F, Guo Y, Wu Q, Luo S, Zhang J, Li H, Hu S, Wu B, Lin G, Qiu H, Niu B, Sun X, Xu L, Lu J, Du X, Wang Z, Wang X, Kang L, Wang Z, Wang Q, Liu Q, Xiao Y. Interaction analysis of high-risk pathological features on adjuvant chemotherapy survival benefit in stage II colon cancer patients: a multi-center, retrospective study. BMC Cancer. 2023 Sep 18;23(1):797. doi: 10.1186/s12885-023-11196-4. PMID 37718392